CLINICAL TRIAL: NCT06569966
Title: The Effects of Colorectal Prehabilitation Via Reinfusion or Retention Enema of Ileal Contents Filtrate on the Defecation Functions for the LAR Patients With Ileostomy Before Stoma Closure: A Single Center Prospective Randomized Controlled Study
Brief Title: The Effects of Colorectal Prehabilitation Via Reinfusion or Retention Enema of Ileal Contents Filtrate on the Defecation Functions for the LAR Patients With Ileostomy Before Stoma Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prehab-LARS2024
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation Group (Experimental): The contents of the ileostomy were collected and placed in a wide mouth container, mixed with 500mL normal temperature saline, and placed in a funnel with double layer medical gauze. The filtrate of the ileal contents was collected and placed into an enema for use. The catheter was placed into the ileal output end of the ostomy through anterograde enema or transanal retention enema, and slowly infused for 15-20 minutes, 2-3 times a day for 4 weeks. The adverse reactions such as abdominal pain, abdominal distension and fever were observed. The number, time, antegrade/retrograde prehabilitation operation, adverse reactions during the operation and other special conditions were recorded every day, and the weight of the patient was recorded.
  Interventions: Behavioral: preoperative prehabilitation treatment of ileostomy contents filtrate reinfusion through distal ileocolon or retention of enema colon
- Perioperative management group (No Intervention): Perioperative management group

INTERVENTIONS:
Behavioral: preoperative prehabilitation treatment of ileostomy contents filtrate reinfusion through distal ileocolon or retention of enema colon — The contents of the ileostomy were collected and placed in a wide mouth container, mixed with 500mL normal temperature saline, and placed in a funnel with double layer medical gauze. The filtrate of the ileal contents was collected and placed into an enema for use. The catheter was placed into the ileal output end of the ostomy through anterograde enema or transanal retention enema, and slowly infused for 15-20 minutes, 2-3 times a day for 4 weeks. The adverse reactions such as abdominal pain, abdominal distension and fever were observed. The number, time, antegrade/retrograde prehabilitation operation, adverse reactions during the operation and other special conditions were recorded every day, and the weight of the patient was recorded
  Arms: Prehabilitation Group

SUMMARY:
This study was a single-center RCT study to compare the effect of preoperative prehabilitation treatment of ileostomy contents filtrate reinfusion through distal ileocolon or retention of enema colon with that of traditional treatment in patients with bowel function after stoma closure.

DETAILED DESCRIPTION:
The patients in the experimental group collected the contents of the ileostomyand placed in a wide mouth container, mixed with 500mL normal temperature saline, and placed in a funnel with double layer medical gauze. The filtrate of the ileal contents was collected and placed into an enema for use. The catheter was placed into the ileal output end of the ostomy through anterograde enema or transanal retention enema, and slowly infused for 15-20 minutes, 2-3 times a day for 4 weeks. The adverse reactions such as abdominal pain, abdominal distension and fever were observed. The number, time, antegrade/retrograde prehabilitation operation, adverse reactions during the operation and other special conditions were recorded every day, and the weight of the patient was recorded.Patients in the control group received routine perioperative management.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-85 years old
* Karnofsky performance status (KPS)≥70%; Or ECOG score 2 points or less
* rectal cancer confirmed by preoperative pathology
* in the rectum resection before low, low colorectal anastomosis or after neoadjuvant therapy of patients
* prophylactic ileostomy.

Exclusion Criteria:

* cannot complete treatment
* the history of the anorectal surgery
* preoperative bowel dysfunction such as diarrhea, irritable bowel syndrome and functional constipation, etc.)
* postoperative anastomotic fistula and stricture
* during pregnancy or breastfeeding women
* with uncontrolled seizures, central nervous system disease or a history of mental disorders
* the last five years have other history of malignant disease cured except skin cancer and cervical carcinoma in situ
* clinically significant (i.e., active) heart disease, such as symptomatic coronary artery disease, New York Heart Association class II or worse 9) severe congestive heart failure or major arrhythmia requiring medical intervention, or myocardial infarction within the previous 6 months
* has a history of cerebral infarction or cerebral hemorrhage within the past 6 months
* organ transplantation requiring immunosuppressive therapy
* serious uncontrolled repeated infections, or other serious with disease of control;
* moderate or severe renal impairment creatinine clearance equal to or less than 50ml/min, or upper limit of normal (ULN)
* emergency surgery due to tumor emergencies (bleeding, perforation, obstruction)
* in screening the first 4 weeks received study medication or treatment (to participate in other test).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The extent of low anterior resection syndrome | 1 month after discharge, and 3, 6, and 12 months after surgery
  low anterior resection syndrome score（0-42，Higher scores indicate more severe symptoms）

SECONDARY OUTCOMES:
the intestinal function recovery | up to 10 days after surgery
  The first postoperative exhaust and defecation time
Concentration of C-reactive protein | up to 10 days after surgery
  Concentration of C-reactive protein after surgery
Quality of Life Questionnaire Core 30 | 1 month after discharge, and 3, 6, and 12 months after surgery
  Quality of Life Questionnaire Core 30（0-100，standardscore，A higher score in the symptom domain indicates a worse quality of life）
fecal incontinence | 1 month after discharge, and 3, 6, and 12 months after surgery
  The Cleveland clinic fecal incontinence score（0-20，Higher scores indicate more severe symptoms）
Weight change after rehabilitation | From date of randomization until the date of stoma closure surgery, assessments usually take up to 3 months
  Weight change after rehabilitation
The number of emergency visits or rehospitalizations related to stoma closure | 1 year after surgery
  The number of emergency visits or rehospitalizations related to stoma closure
the incidence of postoperative intestinal obstruction (POI) | 1 year after surgery
  the incidence of postoperative intestinal obstruction (POI)

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Zhou, Study Chair — the Affiliated Hospital of Qingdao
Locations (1):
- the Affiliated Hospital of Qingdao, Qingdao, Shandong, China